CLINICAL TRIAL: NCT03407235
Title: Laparoscopic Skill Acquisition; Can the Loss of Depth Perception Associated With Laparoscopic Surgery be Adequately Simulated by an Eye Patch?
Brief Title: Simulating Laparoscopy With an Eye Patch
Acronym: LapACQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LTf15082013 ammend. 2
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2017-12

CONDITIONS: Laparoscopic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Novices (Other): Four laparoscopic task will be undertaken on a computerized laparoscopic trainer and box trainer with eye patch.
  Time to completion is recorded.
  Interventions: Device: Computerized Laparoscopic Trainer; Device: Box trainer with eye patch

INTERVENTIONS:
Device: Computerized Laparoscopic Trainer — Gold standard laparoscopic trainer using simulated computerized equipment.
Device: Box trainer with eye patch — Simple, cost effective box trainer, with loss of dept perception achieved with use of eye patch

SUMMARY:
Comparison of laparoscopic training simulator v use of eye patch (to simulate loss of dept perception) to investigate acquisition of laparoscopic skills.

DETAILED DESCRIPTION:
Healthy volunteers who are laparoscopic novices will perform four validated laparoscopic training exercises on both the laparoscopic computerized trainer and on a simple box trainer with an eye patch.

Novices will be allowed to familiarize themselves with the laparoscopic instruments and will be shown short video clips to demonstrate tasks.

They then will have five minutes to complete each of the four tasks. They will return 1-2 weeks later to complete the same process on the alternative training method.

All participants will complete the tasks on both the computerized lap simulator and the box trainer.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic Novices
* 20-40 years
* All genders

Exclusion Criteria:

* Previous laparoscopic surgical experience

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Time to completion of laparoscopic tasks. | 5 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University Of Nottingham, Derby
  - The Medical School, University of Nottingham, Royal Derby Hospital., Derby

IPD SHARING:
Plan to Share IPD: No